CLINICAL TRIAL: NCT00241072
Title: A Single Center, Open Label, Single Arm Trial To Evaluate The Effect Of Twenty Four Weeks Of Treatment With 80 Mg To 320 Mg Valsartan On Insulin Sensitivity In Subjects With Impaired Glucose Tolerance (Igt)
Brief Title: Clinical Trial To Evaluate The Effect Of Valsartan On Insulin Sensitivity In Subjects With Impaired Glucose Tolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489A2412
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension; Impaired Glucose Tolerance
MeSH Terms: conditions — Hypertension; Glucose Intolerance | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan — 24 WEEKS OF TREATMENT WITH VALSARTAN (80 MG - 320 MG)

SUMMARY:
THE PURPOSE OF THIS STUDY IS TO DETERMINE IF 24 WEEKS OF TREATMENT WITH VALSARTAN (80 MG - 320 MG) IMPROVES INSULIN SENSITIVITY IN SUBJECTS WITH HIGHER THAN NORMAL GLUCOSE LEVELS USING A TEST CALLED THE EUGLYCEMIC CLAMP.

ELIGIBILITY:
Inclusion Criteria:

history or presenting hypertension Elevated fasting blood glucose levels -

Exclusion Criteria:

Pregnancy potential Diabetes mellitus

Other criteria apply

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline insulin sensitivity after 24 weeks

SECONDARY OUTCOMES:
Change from baseline in the function of cells that line blood vessels after 24 weeks
Change from baseline in markers of vascular inflammation after 24 weeks
Adverse events and serious adverse events at each study visit for 24 weeks
Hematology, blood chemistries, and urine measurements for up to 24 weeks
Vital signs and physical examinations for up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals